CLINICAL TRIAL: NCT04370249
Title: Construction of a Composite Clinical-echo Score Predictive of a Risk of Short-term Aggravation of Respiratory Impairment in Patients Suspected of Covid-19
Acronym: VIRUS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: WINFOCUS-France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC20_0164
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with suspected COVID-19 infection: Patients admitted and managed in an emergency department under suspicion of COVID-19 infection who received a pleuro-pulmonary ultrasound on admission
  Interventions: Other: pulmonary ultrasound

INTERVENTIONS:
Other: pulmonary ultrasound — pulmonary ultrasound on admission

SUMMARY:
With the influx of patients suspected of Covid-19 and the limited number of hospital beds, there is a need for sensitive triage to detect patients at risk of pulmonary complications and therefore requiring hospitalization, but also specific triage to safely discharge patients without risk factors or signs of clinical or ultrasound severity. The use of pulmonary ultrasound in addition to clinical assessment seems appropriate. Indeed, it allows early detection of signs of pneumopathy which, in the current context, most often correspond to Covid-19. These signs include B-lines, which indicate interstitial pulmonary oedema, and an anfractuous and thickened pleural line, or even centimetric parenchymal condensations with a low level of pleural effusion. Conversely, the presence of a medium to large pleural effusion is not very suggestive of the diagnosis of Covid-19. In addition, a lung ultrasound score has been developed and validated to assess the severity of acute respiratory distress and predict the occurrence of acute respiratory distress syndrome. It is based on the performance of a 12-point (6 per hemi-thorax) pulmonary ultrasound with the collection of the presence of B-lines, condensation or pleural effusion. In the hands of a trained operator, this examination takes only a few minutes.

The aim of the study is to develop a score based on clinical and ultrasound evidence to allow early and safer referral than that based on clinical evidence alone. To do this, the study will retrospectively collect clinical and lung ultrasound data from departments that use this technique on a daily basis.

DETAILED DESCRIPTION:
The objective of the VIRUS research is therefore to develop an innovative clinical-echo score (VIRUScore), based on risk factors, clinical elements and ultrasound data. This predictive score corresponds to a probabilistic measure of the individual risk of aggravation and is intended to become the cornerstone of a decision-making algorithm for triaging/managing COVID-19 patients (VIRUS algorithm). Initial VIRUScore and evolution of clinical and/or clinico-biological signs will thus have to arbitrate different patient pathway scenarios with 2 major objectives: first, to reduce hospital tension and desaturate emergency departments and COVID-19 units to ensure maximum monitoring of moderate forms, some of which are likely to evolve towards severe forms. The negative predictive value of severe short-term aggravation (H48) should therefore be maximized for these patient profiles invited to return home and/or transfer to non-specialized hospitals or clinics. And secondly, it should be sensitive in detecting and predicting the most severe forms with a high risk of resuscitative escalation and/or death, allowing prioritization (access to CT, access to research protocols) and grading the intensity of clinical surveillance, for anticipation of resuscitative resources.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted and managed in an emergency department under suspicion of COVID-19 who received a pleuro-pulmonary ultrasound on admission

Exclusion Criteria:

* Patients admitted and treated in an Emergency Department for suspected COVID-19 but who did not receive a pleuro-pulmonary ultrasound on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for VIRUS corresponds to all patients admitted to Emergency Departments on suspicion of COVID-19 (established by primary care professionals or during regulation by the EMS).
Sampling Method: Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2020-04-09 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Construction of a composite clinical-echo score (VIRUScore) predictive of risk of worsening respiratory impairment in COVID-19 adult patients admitted to the Emergency Department | 48 hours post-admission
  Multivariate model predictive of clinical worsening of respiratory impairment within 48 hours post-admission : intubation, oxygenotherapy, need of vasoactive drugs, worsening of state,age, gender, body surface, LUScore (pulmonary ultrasound), FiO2, need of ventral decubitus, risk factor (obesity, asthma...), time from the beginning of the first symptoms

SECONDARY OUTCOMES:
Evaluate the prognostic performance of the VIRUScore on the risk of pulmonary aggravation | 48 hours post-admission
  Sensitivity, specificity, positive predictive value, negative predictive value of VIRUScore on risk of pulmonary aggravation
Evaluate the prognostic performance of the VIRUScore on the risk of severe pulmonary aggravation defined by resuscitation admission and/or death at D14 (sensitivity, specificity, positive predictive value, negative predictive value). | 14 days post-admission
  Sensitivity, specificity, positive predictive value, negative predictive value of VIRUScore on the risk of severe pulmonary aggravation defined by resuscitation admission and/or death.
Construction of a decisional algorithm for triage and management of COVID-19 patients. | 14 days post-admission
  Research of VIRUScore cut-off values maximizing the negative predictive value and construction of a decisional algorithm maximizing returns home and transfers to non-specialized hospitals or clinics without loss of individual chance.
Search for "ultrasound signature" (lung fields and/or severity of involvement) associated with mild (return home) vs. moderate (oxygen therapy) vs. severe (resuscitation/death) clinical forms. | 14 days post-admission
  Search for "Ultrasound signature" (lung fields and/or severity of damage) associated with mild vs. moderate (oxygen therapy) vs. severe (resuscitation/death) clinical forms.
Evaluate the analytical concordance between the pulmonary ultrasound (LUScore) and the Gold-standard CT-scan (CT score) | 14 days post-admission
  Diagnostic concordance of the LUScore and CT score with the severity grades defined by the French Radiology Society
Construction of a score predictive of aggravation in the sub-population of patients returned home | 14 days post-admission
  Predictive Score for Aggravation in Patients Returned Home

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nantes, Nantes, France